CLINICAL TRIAL: NCT01133197
Title: The Impact of Thumb Carpometacarpal Osteoarthritis on General Health
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Principal Investigator, Ryan Calfee, MD, Associate Professor of Orthopaedic Surgery, Washington University School of Medicine
Other Study IDs: 09-0829
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Thumb Arthritis
Keywords: thumb; arthritis; Impact of thumb arthritis on health
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- controls: No hand arthritis
- CMC Arthritis: Patients with arthritis

SUMMARY:
This study is designed to define the impact of thumb arthritis on patient's general health. As a secondary objective, data will be analyzed to determine the effects of medical and musculoskeletal comorbidities on the rating of upper extremity function by the patient.

DETAILED DESCRIPTION:
This study is designed to define the impact of thumb arthritis on patient's general health. As a secondary objective, data will be analyzed to determine the effects of medical and musculoskeletal comorbidities on the rating of upper extremity function by the patient.

Potential Contribution: The data that we intend to gather could further our understanding of the overall health impact of thumb osteoarthritis and allow surgeons to more accurately interpret patient-rated measures of upper extremity function in the presence of comorbidities.

Osteoarthritis of the thumb carpometacarpal joint is one of the most common sites of arthritic degeneration in the hand. To date, no study has examined this conditions impact on overall health using a validated health measure (e.g. SF-36). Additionally, no study has examined the impact of medical and musculoskeletal comorbidities on patient-rated measures of upper extremity function in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults clinically diagnosed with thumb carpometacarpal osteoarthritis. The diagnosis must have been confirmed radiographically prior to consideration for study enrollment.
* Adults accompanying patients to participating offices will be recruited to be control subjects. They must not be receiving medical or surgical treatment for a hand or wrist complaint.
* Additionally control subjects must not have been diagnosed with thumb osteoarthritis.

Exclusion Criteria:

* Subjects must be over 18 years of age and English speaking.
* Subjects are not to include incarcerated adults or those unable to provide consent for study participation.
* Patients diagnosed with currently symptomatic hand or wrist pathology outside of the thumb carpometacarpal joint will be excluded.
* Patient with prior surgery on the affected thumb will be excluded.
* Pregnant females are excluded from study participation with pregnancy determined by patient self-reporting (standard of care before office radiographs).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting for treatment have thumb arthritis
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2009-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Hand Function | Baseline
  Use of hand by Michigan Hand Questionnaire

SECONDARY OUTCOMES:
Overall Health | Baseline
  SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Ryan P Calfee, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States